CLINICAL TRIAL: NCT00441311
Title: Dissemination of Colorectal Cancer Screening to Primary Care Physicians
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sherri Gorin, PhD, Columbia University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAA6315
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; primary care physicians; health disparities; stratified randomized clinical trial
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Academic Detailing (Experimental): The academic detailing intervention will involve multiple components some of which are standardized across physicians (i.e. self-learning packets, newsletters). Detailing will also be customized to each physician, although the frequency of the detailing visits will be routinized across all participants to reduce cost and to maximize its potential for dissemination.
  Interventions: Behavioral: Academic Detailing
- Service-as-Usual (No Intervention): Control Arm

INTERVENTIONS:
Behavioral: Academic Detailing — The academic detailing intervention will involve multiple components some of which are standardized across physicians (i.e. self-learning packets, newsletters). Detailing will also be customized to each physician, although the frequency of the detailing visits will be routinized across all participants to reduce cost and to maximize its potential for dissemination.
  Arms: Academic Detailing

SUMMARY:
The aim is to assess the efficacy of an intervention, academic detailing, a brief, frequently repeated educational program, on increasing recommendations for colorectal cancer screening among primary care providers by comparison to a service-as-usual control. The study is a stratified randomized clinical trial of primary care physicians, stratified by distinct urban communities in the New York metropolitan area. The primary outcome is colorectal cancer screening recommendations measured via medical audit at 12-month followup after randomization.

DETAILED DESCRIPTION:
The purpose of the present study is to adapt and extend the use of academic detailing to the dissemination of colorectal cancer (CRC) screening findings and guidelines to primary care physicians practicing in selected geographic areas in New York City. Since improving implementation of cancer screening guidelines also involves compliance by patients in completing the recommended tests or examinations, we will also seek to assess knowledge, attitude and screening behaviors of patients visiting primary care practitioners in our sample. Our long-term goal is to reduce colorectal cancer mortality among ethnic and racial minorities, by influencing the screening behaviors of their primary care physicians.

The specific aims of the study are as follows:

* Aim 1. To test the hypothesis that an intervention, multi-component academic detailing, will increase the rate of physician CRC screening at 3and 6month postrandomization, compared to the rate observed in a serviceasusual control.
* Aim 2. To develop models predicting which physician offices are most and least likely to adopt the intervention, and to generate hypotheses about tailoring the dissemination of CRC screening guidelines to different physician subgroups.
* Aim 3. To conduct cost-effectiveness analysis comparing the incremental societal costs and effects (in lives saved, life-years saved, and quality-of-life-years saved) of the CRC intervention implemented in physicians' offices.

ELIGIBILITY:
Inclusion Criteria:

* Devote at least 50% of their practice to primary care
* Work in the study communities
* Are non-hospital based community practitioners
* Have no immediate plans to retire or to leave their practice.

Exclusion Criteria:

* Specialty physicians
* Intend to retire or otherwise leave practice over course of the study
* Other conditions that would preclude meaningful participation
* Not working in study communities

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2003-05; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening recommendations | Up to 12 months from the time of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Sheinfeld Gorin, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Honda K, Gorin SS. A model of stage of change to recommend colonoscopy among urban primary care physicians. Health Psychol. 2006 Jan;25(1):65-73. doi: 10.1037/0278-6133.25.1.65. PMID 16448299